CLINICAL TRIAL: NCT05530681
Title: Correlation Pelvic Floor Function and Ultrasound Findings One Year After Childbirth
Acronym: DeliverUU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: s66245
Record Dates: First submitted 2022-07-06; First posted 2022-09-07 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Pelvic Floor Disorders; Obstetric Trauma; Urinary Incontinence; Anal Incontinence; Pelvic Organ Prolapse; Pelvic Pain; Sexual Dysfunction; Constipation; Anal Sphincter Injury
Keywords: urinary incontinence; anal incontinence; pelvic organ prolapse; sexual dysfunction; constipation; postpartum; levator avulsion; anal sphincter injury
MeSH Terms: conditions — Pelvic Floor Disorders; Urinary Incontinence; Encopresis; Pelvic Organ Prolapse; Pelvic Pain; Sexual Dysfunction, Physiological; Constipation | interventions — Pain Measurement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental)
  Interventions: Diagnostic Test: Questionnaire; Diagnostic Test: Pelvic floor ultrasound

INTERVENTIONS:
Diagnostic Test: Questionnaire — The survey consists in standardized and validated questionnaires on urinary function (ICIQ-SF, 4 items), bowel function (SMIS, 7 items and PAC-SYM, 12 items), symptoms of prolapse (POPDI, 6 items) and sexual function (Female Sexual Function Index FSFI, 19 items and Female Sexual Distress Scale - Revised FSDS-R, 13 items). questionnaire will be used at recruitment, at the postpartum visit, at the first annual follow-up visit.
Diagnostic Test: Pelvic floor ultrasound — Pelvic floor ultrasound is the preferred imaging modality for documenting pelvic floor anatomy during pregnancy or after delivery. This examination is routinely performed in the outpatient clinic during patient visits (including the one year check-up after delivery). The technique used to assess the pelvic floor is described in detail in the 2019 practice parameters issued by IUGA.
  Other Names: Transperineal ultrasound; Pelvic floor sonography

SUMMARY:
This is a single-center prospective cohort study sponsored by the University Hospitals Leuven (UZ). Women will undergo a pelvic floor ultrasound and will be asked to fill out a questionnaire at the time of their admission into the labour suite, at the postpartum check-up and 12 months postpartum.

The primary objective is to correlate self-reported symptoms of Pelvic Floor Dysfunction (PFD) (binary outcome) at one year after delivery with structural changes to the Pelvic Floor Muscles (PFM) and postpartum evidence of levator avulsion (binary indicator) as measured by TransPerineal UltraSound (TPUS).

Secondary objectives are to compare demographical and obstetrical variables between patients suffering from PFD symptoms or pelvic floor injury (documented one year after delivery) and those who do not; to record how patients manage and cope with PFD including recovery and compliance with Pelvic Floor Muscle Training (PFMT) as prescribed in the standard pathway of peripartum care; and to use of TPUS images for the development of artificial intelligence tools for automated image analysis.

Primary outcomes are PFD symptoms one year after delivery and injury to the PFM evidenced by POP-Q and TPUS. The demographic variables and information about the pregnancy and the delivery will be obtained from the medical records.

The presence and severity of PFD will be measured using standardized self-reporting tools: Pelvic Organ Prolapse Distress Index (POP-DI), Patient Assessment Constipation-SYMptoms (PAC-SYM), International Consultation on Incontinence Questionnaire - Urinary Incontinence - Short Form (ICIQ-SF), St. Mark's Incontinence Score (SMIS), Female Sexual Function Index (FSFI), Female Sexual Distress Scale - Revised (FSDS-R). FSFI is a widely used generic tool with sufficient granularity and validated in a large number of languages. FSDS-R assesses the construct "personal distress", which has been considered as an additional important aspect contributing to sexual dysfunction of women.

PFD, as a clustered outcome, being the presence of any kind of pelvic floor dysfunction symptoms, will be defined as POP-DI score of ≥11 OR ICIQ-SF score of ≥1 OR SMIS score of ≥1 OR FSFI score ≤ 26.55 OR FSDS-R score ≥11.

ELIGIBILITY:
Inclusion Criteria:

* age = or > 18 years
* Dutch/English-speaking
* > 33 weeks gestation
* delivering in UZ Leuven
* vaginal delivery

Exclusion Criteria:

* age < 18 years
* not Dutch/English-speaking
* < 33 weeks gestation
* not delivering in UZ Leuven
* non-vaginal delivery
* Any disorder, that independently from delivery, affects pelvic floor function or structure, such as, but not limited to musculoskeletal or neurologic diseases.
* any women with drug addiction, cognitive deficit, language-barrier and illiteracy
* any disorder or timing or circumstances, which in the Investigator's opinion represents an obstacle to proper informed consent, or safe and/or compliant participation.
* any prior or simultaneous treatment(s) potentially jeopardising safety or compromising trial integrity.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 320 (Estimated)
Dates: Start 2022-08-17 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Urinary incontinence | one year postpartum
  International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-SF) score of ≥1 (score range 0-21, higher scores mean worse urinary incontinence)
Anal Incontinence | one year postpartum
  St Mark's Incontinence Score (SMIS) ≥1 (score range 0-24, higher scores mean worse anal incontinence)
Sexual dysfunction | one year postpartum
  Female Sexual Function Index (FSFI) score ≤ 26.55 (score range 2 to 36, worse scores mean worse sexual function) OR FSDS-R score ≥11 (score range 0 to 52, with higher scores indicating more sexually related distress)
Constipation according to the Rome IV criteria | one year postpartum
  Must include two or more of the following:** Straining during more than ¼ (25%) of defecations Lumpy or hard stools (Bristol Stool Form Scale 1-2) more than ¼ (25%) of defecations Sensation of incomplete evacuation more than ¼ (25%) of defecations Sensation of anorectal obstruction/blockage more than ¼ (25%) of defecations Manual maneuvers to facilitate more than ¼ (25%) of defecations (e.g., digital evacuation, support of the pelvic floor) Fewer than three SBM per week Loose stools are rarely present without the use of laxatives Insufficient criteria for irritable bowel syndrome

SECONDARY OUTCOMES:
levator avulsion | 1 year
  complete avulsion is defined as complete detachment of the puborectalis part of the levator ani muscle from the inferior pubic ramus on 3 out of 8 tomographic ultrasound imaging slices of the pelvic floor during contraction
levator hiatus antero-posterior diameter (cm) | 1 year
levator hiatus latero-lateral diameter (cm) | 1 year
levator hiatus surface (cm2) | 1 year
anal sphincter injury | 1 year
  residual defect of at least 30 degrees on Tomographic Ultrasound Imaging
co-contraction | 1 year
  approximation of the dorsal puborectalis to the symphysis pubis during Valsalva manoeuvre
pelvic organ descent | 1 year
  descent of bladder/cervix/ampulla rectalis under the level of the symphysis pubis
bladder neck mobility | 1 year
  axial descent of the bladder neck during Valsalva manoeuvre

CONTACTS AND LOCATIONS:
Overall Officials: Jan Deprest, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZLeuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Avery K, Donovan J, Peters TJ, Shaw C, Gotoh M, Abrams P. ICIQ: a brief and robust measure for evaluating the symptoms and impact of urinary incontinence. Neurourol Urodyn. 2004;23(4):322-30. doi: 10.1002/nau.20041. PMID 15227649
- [Background] Basson R, Berman J, Burnett A, Derogatis L, Ferguson D, Fourcroy J, Goldstein I, Graziottin A, Heiman J, Laan E, Leiblum S, Padma-Nathan H, Rosen R, Segraves K, Segraves RT, Shabsigh R, Sipski M, Wagner G, Whipple B. Report of the international consensus development conference on female sexual dysfunction: definitions and classifications. J Urol. 2000 Mar;163(3):888-93. PMID 10688001
- [Background] Baser RE, Li Y, Carter J. Psychometric validation of the Female Sexual Function Index (FSFI) in cancer survivors. Cancer. 2012 Sep 15;118(18):4606-18. doi: 10.1002/cncr.26739. Epub 2012 Feb 22. PMID 22359250
- [Background] Bo K. Does pelvic floor muscle training prevent and treat urinary and fecal incontinence in pregnancy? Nat Clin Pract Urol. 2009 Mar;6(3):122-3. doi: 10.1038/ncpuro1313. Epub 2009 Feb 3. PMID 19190594
- [Background] Bo K. Pelvic floor muscle training in treatment of female stress urinary incontinence, pelvic organ prolapse and sexual dysfunction. World J Urol. 2012 Aug;30(4):437-43. doi: 10.1007/s00345-011-0779-8. Epub 2011 Oct 9. PMID 21984473
- [Background] Bo K, Braekken IH, Majida M, Engh ME. Constriction of the levator hiatus during instruction of pelvic floor or transversus abdominis contraction: a 4D ultrasound study. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Jan;20(1):27-32. doi: 10.1007/s00192-008-0719-3. Epub 2008 Sep 20. PMID 18806912
- [Background] Bo K, Finckenhagen HB. Vaginal palpation of pelvic floor muscle strength: inter-test reproducibility and comparison between palpation and vaginal squeeze pressure. Acta Obstet Gynecol Scand. 2001 Oct;80(10):883-7. doi: 10.1034/j.1600-0412.2001.801003.x. PMID 11580731
- [Background] Bump RC, Mattiasson A, Bo K, Brubaker LP, DeLancey JO, Klarskov P, Shull BL, Smith AR. The standardization of terminology of female pelvic organ prolapse and pelvic floor dysfunction. Am J Obstet Gynecol. 1996 Jul;175(1):10-7. doi: 10.1016/s0002-9378(96)70243-0. PMID 8694033
- [Background] Callewaert G, Albersen M, Janssen K, Damaser MS, Van Mieghem T, van der Vaart CH, Deprest J. The impact of vaginal delivery on pelvic floor function - delivery as a time point for secondary prevention. BJOG. 2016 Apr;123(5):678-81. doi: 10.1111/1471-0528.13505. Epub 2015 Jul 6. No abstract available. PMID 26147210
- [Background] DeLancey JO. The hidden epidemic of pelvic floor dysfunction: achievable goals for improved prevention and treatment. Am J Obstet Gynecol. 2005 May;192(5):1488-95. doi: 10.1016/j.ajog.2005.02.028. PMID 15902147
- [Background] Derogatis L, Clayton A, Lewis-D'Agostino D, Wunderlich G, Fu Y. Validation of the female sexual distress scale-revised for assessing distress in women with hypoactive sexual desire disorder. J Sex Med. 2008 Feb;5(2):357-64. doi: 10.1111/j.1743-6109.2007.00672.x. Epub 2007 Nov 27. PMID 18042215
- [Background] Dietz HP. Pelvic floor ultrasound: a review. Am J Obstet Gynecol. 2010 Apr;202(4):321-34. doi: 10.1016/j.ajog.2009.08.018. PMID 20350640
- [Background] Dietz HP, Shek C, Clarke B. Biometry of the pubovisceral muscle and levator hiatus by three-dimensional pelvic floor ultrasound. Ultrasound Obstet Gynecol. 2005 Jun;25(6):580-5. doi: 10.1002/uog.1899. PMID 15883982
- [Background] Fleiss JL, Tytun A, Ury HK. A simple approximation for calculating sample sizes for comparing independent proportions. Biometrics. 1980 Jun;36(2):343-6. PMID 26625475
- [Background] Frank L, Kleinman L, Farup C, Taylor L, Miner P Jr. Psychometric validation of a constipation symptom assessment questionnaire. Scand J Gastroenterol. 1999 Sep;34(9):870-7. doi: 10.1080/003655299750025327. PMID 10522604
- [Background] Frawley HC, Galea MP, Phillips BA, Sherburn M, Bo K. Effect of test position on pelvic floor muscle assessment. Int Urogynecol J Pelvic Floor Dysfunct. 2006 Jun;17(4):365-71. doi: 10.1007/s00192-005-0016-3. Epub 2005 Oct 5. PMID 16205845
- [Background] Garcia-Mejido JA, Idoia-Valero I, Aguilar-Galvez IM, Borrero Gonzalez C, Fernandez-Palacin A, Sainz JA. Association between sexual dysfunction and avulsion of the levator ani muscle after instrumental vaginal delivery. Acta Obstet Gynecol Scand. 2020 Sep;99(9):1246-1252. doi: 10.1111/aogs.13852. Epub 2020 Apr 12. PMID 32198764
- [Background] AIUM/IUGA practice parameter for the performance of Urogynecological ultrasound examinations : Developed in collaboration with the ACR, the AUGS, the AUA, and the SRU. Int Urogynecol J. 2019 Sep;30(9):1389-1400. doi: 10.1007/s00192-019-03954-5. No abstract available. PMID 31111173
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Int Urogynecol J. 2010 Jan;21(1):5-26. doi: 10.1007/s00192-009-0976-9. Epub 2009 Nov 25. PMID 19937315
- [Background] Kamel R, Montaguti E, Nicolaides KH, Soliman M, Dodaro MG, Negm S, Pilu G, Momtaz M, Youssef A. Contraction of the levator ani muscle during Valsalva maneuver (coactivation) is associated with a longer active second stage of labor in nulliparous women undergoing induction of labor. Am J Obstet Gynecol. 2019 Feb;220(2):189.e1-189.e8. doi: 10.1016/j.ajog.2018.10.013. Epub 2018 Oct 12. PMID 30321525
- [Background] Madhu C, Swift S, Moloney-Geany S, Drake MJ. How to use the Pelvic Organ Prolapse Quantification (POP-Q) system? Neurourol Urodyn. 2018 Aug;37(S6):S39-S43. doi: 10.1002/nau.23740. PMID 30614056
- [Background] Neijenhuijs KI, Hooghiemstra N, Holtmaat K, Aaronson NK, Groenvold M, Holzner B, Terwee CB, Cuijpers P, Verdonck-de Leeuw IM. The Female Sexual Function Index (FSFI)-A Systematic Review of Measurement Properties. J Sex Med. 2019 May;16(5):640-660. doi: 10.1016/j.jsxm.2019.03.001. Epub 2019 Apr 5. PMID 30956110
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Background] Rostaminia G, Javadian P, Awad C, Shobeiri SA. Ultrasound Indicators of Rectal Support Defect in Women With Obstructive Defecatory Symptoms. Female Pelvic Med Reconstr Surg. 2019 May/Jun;25(3):222-225. doi: 10.1097/SPV.0000000000000511. PMID 29300257
- [Background] Solans-Domenech M, Sanchez E, Espuna-Pons M; Pelvic Floor Research Group (Grup de Recerca del Sol Pelvia; GRESP). Urinary and anal incontinence during pregnancy and postpartum: incidence, severity, and risk factors. Obstet Gynecol. 2010 Mar;115(3):618-628. doi: 10.1097/AOG.0b013e3181d04dff. PMID 20177295
- [Background] ter Kuile MM, Brauer M, Laan E. The Female Sexual Function Index (FSFI) and the Female Sexual Distress Scale (FSDS): psychometric properties within a Dutch population. J Sex Marital Ther. 2006 Jul-Sep;32(4):289-304. doi: 10.1080/00926230600666261. PMID 16709550
- [Background] Thom DH, Rortveit G. Prevalence of postpartum urinary incontinence: a systematic review. Acta Obstet Gynecol Scand. 2010 Dec;89(12):1511-22. doi: 10.3109/00016349.2010.526188. Epub 2010 Nov 5. PMID 21050146
- [Background] Thomas V, Shek KL, Guzman Rojas R, Dietz HP. Temporal latency between pelvic floor trauma and presentation for prolapse surgery: a retrospective observational study. Int Urogynecol J. 2015 Aug;26(8):1185-9. doi: 10.1007/s00192-015-2677-x. Epub 2015 Apr 3. PMID 25837351
- [Background] Urbankova I, Grohregin K, Hanacek J, Krcmar M, Feyereisl J, Deprest J, Krofta L. The effect of the first vaginal birth on pelvic floor anatomy and dysfunction. Int Urogynecol J. 2019 Oct;30(10):1689-1696. doi: 10.1007/s00192-019-04044-2. Epub 2019 Jul 20. PMID 31327032
- [Background] Utomo E, Blok BF, Steensma AB, Korfage IJ. Validation of the Pelvic Floor Distress Inventory (PFDI-20) and Pelvic Floor Impact Questionnaire (PFIQ-7) in a Dutch population. Int Urogynecol J. 2014 Apr;25(4):531-44. doi: 10.1007/s00192-013-2263-z. Epub 2014 Jan 21. PMID 24445668
- [Background] Vaizey CJ, Carapeti E, Cahill JA, Kamm MA. Prospective comparison of faecal incontinence grading systems. Gut. 1999 Jan;44(1):77-80. doi: 10.1136/gut.44.1.77. PMID 9862829
- [Background] van Delft KW, Thakar R, Sultan AH, IntHout J, Kluivers KB. The natural history of levator avulsion one year following childbirth: a prospective study. BJOG. 2015 Aug;122(9):1266-73. doi: 10.1111/1471-0528.13223. Epub 2014 Dec 17. PMID 25514994
- [Background] Wang X, Ji X. Sample Size Estimation in Clinical Research: From Randomized Controlled Trials to Observational Studies. Chest. 2020 Jul;158(1S):S12-S20. doi: 10.1016/j.chest.2020.03.010. PMID 32658647